CLINICAL TRIAL: NCT00640900
Title: A Multi-Site Randomized Trial of a Commercial Weight Loss Program
Brief Title: Food, Activity and Behavior Trial
Acronym: FAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jenny Craig, Inc. (Industry)
Responsible Party: Dr. Cheryl Rock, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20073396
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; weight loss; commercial weight loss program
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Commercial program at center (Experimental)
  Interventions: Behavioral: Commercial weight loss program
- Commercial program over the telephone (Experimental)
  Interventions: Behavioral: Commercial weight loss program
- Usual care (Other): Weight loss counseling
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Usual care — Two individualized weight loss counseling sessions with a dietetics professional, and monthly contacts to maintain communications.
  Arms: Usual care
Behavioral: Commercial weight loss program — Active weekly participation until weight loss goals are reached, and monthly participation to maintain the weight loss.
  Arms: Commercial program at center; Commercial program over the telephone

SUMMARY:
This study will provide data on the response over 24 months to two commercial weight loss programs (center-based and telephone-based) compared to control conditions.

DETAILED DESCRIPTION:
The first study aim is to test, in a randomized controlled trial, whether participation in the multifaceted traditional center-based commercial weight loss intervention program and/or the telephone-delivered commerical program is associated with a greater degree of weight loss at six, 12, and 18 months and whether weight loss is maintained over a 24-month period in overweight or obese women, compared to usual care or control conditions. This study utilizes a randomized study design with subjects assigned to the center-based weight loss program, telephone-delivered program, or a usual care control group. The second study aim is to describe the effect of participation in the weight loss programs (versus control conditions) on circulating lipids (fasting total plasma cholesterol and triglycerides, low-density lipoprotein [LDL] cholesterol, and high-density lipoprotein [HDL] cholesterol), carotenoids (a biomarker of vegetable and fruit intake), insulin, glucose, leptin, C-reactive protein, and vitamin D, and cardiopulmonary fitness. The center-based intervention involves in-person counseling and obtaining food items from the center, whereas the telephone-delivered program involves telephone counseling with food delivered to the home every two weeks.

Secondary aims of this study involve describing the characteristics associated with greater weight loss and maintenance in each of the two intervention arms. The hypothesis to be tested is that selected participant characteristics, such as older or younger age, might be differentially associated with greater success across the two types of programs and approaches.

Notably, the results of this study would contribute valuable data to the scientific knowledge base regarding the various modalities of communication for behavioral interventions (in-person versus telephone counseling). This is an important issue currently being considered and debated among clinical and community-based behavioral and nutritional scientists whose intervention efforts focus on promoting behavior change and positive effects on health-related outcomes such as weight reduction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Initial BMI >25.0 kg/m2 and <40 kg/m2
* A minimum of 15 kg over ideal weight as defined by the 1983 Metropolitan Life Insurance tables
* Willing and able to participate in clinic visits and JC facility interactions at specified intervals and to maintain contact with the investigators for 24 months
* Willing to allow blood collections
* Capable of performing a simple test for assessing cardiopulmonary fitness

Exclusion Criteria:

* Inability to participate in physical activity because of severe disability (e.g., severe arthritic conditions)
* A history or presence of a comorbid diseases for which diet modification and increased physical activity may be contraindicated
* Self-reported pregnancy or breastfeeding or planning a pregnancy within the next two years
* Currently actively involved in another diet intervention study or organized weight loss program
* Having a history or presence of a significant psychiatric disorder or any other condition that, in the investigator's judgment, would interfere with participation in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
weight loss | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Rock, PhD, RD, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Dow CA, Thomson CA, Flatt SW, Sherwood NE, Pakiz B, Rock CL. Predictors of improvement in cardiometabolic risk factors with weight loss in women. J Am Heart Assoc. 2013 Dec 18;2(6):e000152. doi: 10.1161/JAHA.113.000152. PMID 24351700
- [Derived] Thomson CA, Morrow KL, Flatt SW, Wertheim BC, Perfect MM, Ravia JJ, Sherwood NE, Karanja N, Rock CL. Relationship between sleep quality and quantity and weight loss in women participating in a weight-loss intervention trial. Obesity (Silver Spring). 2012 Jul;20(7):1419-25. doi: 10.1038/oby.2012.62. Epub 2012 Mar 8. PMID 22402738
- [Derived] Rock CL, Emond JA, Flatt SW, Heath DD, Karanja N, Pakiz B, Sherwood NE, Thomson CA. Weight loss is associated with increased serum 25-hydroxyvitamin D in overweight or obese women. Obesity (Silver Spring). 2012 Nov;20(11):2296-301. doi: 10.1038/oby.2012.57. Epub 2012 Mar 8. PMID 22402737
- [Derived] Rock CL, Flatt SW, Sherwood NE, Karanja N, Pakiz B, Thomson CA. Effect of a free prepared meal and incentivized weight loss program on weight loss and weight loss maintenance in obese and overweight women: a randomized controlled trial. JAMA. 2010 Oct 27;304(16):1803-10. doi: 10.1001/jama.2010.1503. Epub 2010 Oct 9. PMID 20935338